CLINICAL TRIAL: NCT01060852
Title: Randomized Controlled Trial Efficacy Study of a Media Literacy Education Substance Use Prevention Program for Elementary School-Aged Children
Brief Title: Evaluation of the Media Detective Program for Elementary School-Aged Children to Prevention Substance Use
Acronym: MD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Principal Investigator, Janis Kupersmidt, Senior Research Scientist, Innovation Research & Training
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44DA016044 (NIH)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol Drinking; Tobacco Smoking
MeSH Terms: conditions — Alcohol Drinking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Media Detective (Experimental): 10-lesson elementary school, substance use prevention program developed based upon the Message Interpretation Processing model designed to increase children's critical thinking skills about media messages and reduce intent to use tobacco and alcohol products.
  Interventions: Behavioral: Media Detective

INTERVENTIONS:
Behavioral: Media Detective — 10-lesson elementary school, media literacy education, substance use prevention program. Each lesson takes approximately 45 minutes to teach and was taught every school day for 2 weeks.
  Other Names: Media literacy education

SUMMARY:
The purpose of this study was to determine whether a media literacy education program taught be teacher to late elementary school students (grades 3-5) positively affected students' critical thinking skills and substance use-related health outcomes.

DETAILED DESCRIPTION:
Media Detective is a 10-lesson elementary school, substance abuse prevention program developed based upon the Message Interpretation Processing model designed to increase children's critical thinking skills about media messages and reduce intent to use tobacco and alcohol products. The purpose of this study was to conduct a short-term randomized controlled trial study to evaluate the effectiveness of Media Detective for achieving these goals.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and write in English

Exclusion Criteria:

* None

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 679 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Intent to alcohol or tobacco products | 2 weeks: pretest and posttest

SECONDARY OUTCOMES:
Understanding of the persuasive intent of advertising | 2 weeks: pretest and posttest
Media deconstruction skills | 2 weeks: pretest and posttest
Interest in alcohol-branded merchandise | 2 weeks: pretest and posttest
Self-efficacy to refuse offers to use alcohol or tobacco products | 2 weeks: pretest and posttest

CONTACTS AND LOCATIONS:
Overall Officials: Janis B Kupersmidt, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

REFERENCES:
- See also: innovation Research & Training company website — http://www.irtinc.us